CLINICAL TRIAL: NCT00285740
Title: Group Cognitive Behavioral Therapy to Treat Depression in an Epilepsy Clinic Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Epilepsy Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2903; 34121
Record Dates: First submitted 2006-01-31; First posted 2006-02-02 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Epilepsy; Depressive Disorder
MeSH Terms: conditions — Epilepsy; Depressive Disorder | interventions — Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy (CBT) in a Group Format

SUMMARY:
This study involves a form of group therapy called Cognitive Behavioral Therapy or CBT for depressed patients with Epilepsy. The CBT groups will be tailored for an epilepsy clinic population. There are 12 sessions of therapy in the study held once a week for 12 weeks.

DETAILED DESCRIPTION:
Depression is frequent in PWE and often missed for unclear reasons. Busy neurology clinics and their overworked physicians often lack psychiatric backup that may make inquiring about psychological issues problematic. In the psychiatric community, awareness of the need for depression intervention in the primary care clinic has been recognized for many years and several treatment models exist. This study will attempt to use one such model, i.e. Cognitive-Behavioral Therapy (CBT) using a group format and tailoring its use for an epilepsy clinic population.

ELIGIBILITY:
Inclusion Criteria::- Patients will be screened with the Beck Depression Inventory. Those reaching the positive cut-off score of 11 (indicating at least a mild depression) will be entered into the study. Patients entered on antidepressants will be held at a stable dosage. Anti-epileptic drugs will also be maintained on the same dosage at entry into the study when possible clinically, after consultation with their neurologist. Exclusion Criteria:- Patients will be excluded if there is any active serious medical conditions, Standard Score<70 as assessed via the Wide Range Achievement Test, psychotic or substance abuse issues, those who are unable to maintain a stable dose of medications for the duration of study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2005-08 (Actual); Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory

SECONDARY OUTCOMES:
NDDI

CONTACTS AND LOCATIONS:
Overall Officials: John J Barry, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States